CLINICAL TRIAL: NCT06915987
Title: Exercise Snacks for People With Parkinson Disease: A Pilot Randomized Controlled Trial
Brief Title: Parkinson Disease and Exercise Snacks
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Daryl Wile, Clinical Investigator, UBC Southern Medical Program CCDPM Clinical Associate Professor, UBC Dept. Medicine, Div. Neurology, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: H24-02753
Record Dates: First submitted 2025-03-14; First posted 2025-04-08 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Exercise Snacks; Exercise Intervention
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Snack (Active Comparator): Participants to receive higher intensity exercise snack exercises
  Interventions: Behavioral: Exercise Intervention
- Active Movement Breaks (Placebo Comparator): While not a true placebo (i.e., no intervention at all) participants in this arm will receive low intensity / stretching based exercises throughout the study period.
  Interventions: Behavioral: Exercise Intervention

INTERVENTIONS:
Behavioral: Exercise Intervention — Exercise snack group will be higher intensity movements designed to elevate heart rate while active movement break will have low intensity / stretching exercises assigned to them.
  Other Names: Movement Breaks

SUMMARY:
People with Parkinson's Disease (PD) benefit from exercise, but many face barriers like motor disability, fatigue, and lack of time, leading to reduced activity. This study aims to assess the effectiveness of "exercise snacks," short bursts of vigorous activity that can be done anywhere without equipment or a significant time commitment. These exercise snacks help integrate activity into daily life, making it more accessible for people with PD. The secondary goal is to evaluate the feasibility of this approach through this pilot randomized controlled trial (RCT) to inform a larger, future RCT.

DETAILED DESCRIPTION:
Exercise has increasingly become a recognized and valuable component of treatment for individuals with Parkinson's Disease (PD). Numerous studies indicate that exercise can improve motor symptoms, enhance mobility, and contribute to overall well-being. However, despite the well-documented benefits, a significant proportion of people with PD remain inactive. Their physical activity levels often decline over time due to a range of disease-related and practical barriers.

Disease-specific challenges may include motor impairments, fatigue, and apathy. Practical obstacles such as limited time, lack of access to appropriate facilities or programs, adverse weather conditions, and financial constraints also hinder participation. These barriers are compounded in rural and remote communities where exercise resources are scarce. Consequently, there is a pressing need for time-efficient, accessible exercise options adaptable to different stages of PD and feasible for those with varying levels of motor impairment.

Our proposal introduces an innovative intervention called "exercise snacks," consisting of brief, vigorous activity bursts that can be performed anywhere without specialized equipment or a significant time commitment. This approach integrates exercise into daily routines, making it a practical and accessible option for people with PD. Short bouts of exercise are more likely to be maintained and are perceived as more manageable than traditional long-duration workouts. Moreover, this intervention aligns with the World Health Organization Guidelines on Physical Activity and Sedentary Behavior and the Canadian 24-Hour Movement Guidelines for Adults, which encourage breaking up sedentary behavior with short activity breaks.

Exercise interventions must be inclusive to benefit a broader range of people with PD. Many existing studies exclude participants with mild cognitive impairment or those who require assistance with walking or daily activities. Our intervention is specifically designed to accommodate a wide range of abilities. With remote delivery through the Seven Movements platform, the intervention can reach participants in rural or remote areas, where access to traditional exercise programs is limited. This is particularly beneficial in the Interior of British Columbia, where a higher proportion of rural residents face significant healthcare disparities.

Evidence from other populations suggests that exercise snacks can significantly improve cardiovascular fitness and overall health outcomes. High-intensity interval training (HIIT) and similar time-efficient exercise programs have demonstrated comparable benefits to longer-duration aerobic training. We theorize that exercise snacks will offer similar advantages for people with PD by enhancing walking performance, reducing fear of falling, and improving quality of life.

This is an unblinded, block-randomized parallel-group clinical trial involving 40 male and female adults with clinically established PD. Participants will be recruited from Kelowna, British Columbia, through the Humphrey's Family Movement Disorder Clinic and local PD patient support groups. The trial aims to be inclusive, ensuring that the interventions are safe and accessible for a diverse participant population.

Participants with a clinical diagnosis of Parkinson Disease will be randomized to Exercise Snack or Active Movement breaks. Specific hypotheses are: 1) participants in the Exercise Snacks and Active Movement Break groups will be highly adherent to the prescribed activity and 2) people with PD randomized to the Exercise Snacks group will experience improvements in walking performance, reduced fear of falling, and enhanced quality of life compared to the Active Movement Breaks group.

Estimates of the effect of either randomized group assignment includes 1) functional mobility measures (Timed Up and Go, walking speed, balance scales) and 2) psychosocial measures (psychological well-being, fear of falling, quality of life). These will be assessed pre- and post- intervention.

Overall objectives to the study include:

1. to conduct a 12-week pilot randomized controlled trial (RCT) comparing Exercise Snacks to a placebo exercise intervention (Active Movement Breaks) in people with PD
2. measure changes in patient-reported activity levels, fear of falling, quality of life, and clinical measures of walking performance and balance
3. evaluate feasibility outcomes to guide scalability for a fully powered RCT
4. identify barriers and facilitators for exercise snacks in PD patient population using participant-orientated, qualitative study review
5. determine eligibility, recruitment, adherence, and dropout rates for a study of this design

This comprehensive Snack PD pilot design will provide robust evidence on the feasibility and efficacy of exercise snacks for people with PD, informing future large-scale trials and broader implementation strategies.

ELIGIBILITY:
Inclusion Criteria:

* Adults (19 years of age or older) with Clinically Established PD (Postuma et al., 2015).
* Medically cleared to exercise by their physician.
* A score of ≤3 on the modified Hoehn & Yahr scale (i.e. physically independent, may have unilateral or bilateral clinical signs, including mild impairment of postural reflexes).
* Have access to a computer, tablet, or smartphone with internet connection for intervention delivery and tracking.

Exclusion criteria

* Comorbid condition with physical disability preventing participation in exercise (i.e., that cannot be accommodated with modifications to the prescribed exercise).
* A score of >=4 on the modified Hoehn & Yahr scale (meaning they may be able to stand or walk but are not physically independent; this typically includes a need for gait aids such as a cane or walker)
* No access to reliable internet connection.
* Are currently participating in another clinical trial that would interfere with the study procedures described.
* Have a scheduled event (e.g. medical or surgical procedure, prolonged travel in the next 3-4 months) that would interrupt participation in the study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Intervention: completion rate | 10 weeks
  Feasibility of the study intervention by using quantitative data from activities logged in the Seven Movements platform is a primary outcome. The investigators will evaluate this outcome measure of feasibility by looking at multiple variables indicating completion of target exercise. One of the variables used to assess this primary outcome measure of feasibility is activities completion rate of at least 2 sessions five days per week, or 10 per week long block. Threshold values are High (>70%), moderate (50-69%), or low (<50%) adherence. This data will be extracted from the 7 Movements App.
Feasibility of Intervention: rate of perceived exertion | 10 weeks
  Feasibility of the study intervention by using quantitative data from activities logged in the Seven Movements platform is a primary outcome. The investigators will evaluate this outcome measure of feasibility by looking at multiple variables indicating completion of target exercise. One of the variables used to assess this primary outcome measure of feasibility is the intensity of the exercise expecting a rate of perceived exertion (RPE) of >4/10 on the Borg CR-10 scale for Exercise Snacks. This data will be extracted from the 7 Movements App.
Feasibility of Intervention: exercise enjoyment scale | 10 weeks
  Feasibility of the study intervention by using quantitative data from activities logged in the Seven Movements platform is a primary outcome. The investigators will evaluate this outcome measure of feasibility by looking at multiple variables indicating completion of target exercise. One of the variables used to assess this primary outcome measure of feasibility a summary of the Exercise Enjoyment Scale ratings of exercises to compare the study groups. This quantitative data will be extracted from the 7 Movements App.
Adherence to the Intervention: completion rate | 10 weeks
  Adherence of the study intervention will be evaluated using quantitative data from activities logged in the Seven Movements platform is a primary outcome. The investigators will evaluate this outcome measure of adherence by looking at multiple variables indicating completion of target exercise. One of the variables used to assess this primary outcome measure of adherence is activities completion rate of at least 2 sessions five days per week, or 10 per week long block. Threshold values are High (>70%), moderate (50-69%), or low (<50%) adherence. This data will be extracted from the 7 Movements App.
Adherence to the Intervention: rate of perceived exertion | 10 weeks
  Adherence of the study intervention by using quantitative data from activities logged in the Seven Movements platform is a primary outcome. The investigators will evaluate this outcome measure by looking at multiple variables indicating completion of target exercise. One of the variables used to assess this outcome measure of adherence is the intensity of the exercise expecting a rate of perceived exertion (RPE) of >4/10 on the Borg CR-10 scale for Exercise Snacks. This data will be extracted from the 7 Movements App.
Adherence to the Intervention: exercise enjoyment scale | 10 weeks
  Adherence of the study intervention by using quantitative data from activities logged in the Seven Movements platform is a primary outcome. The investigators will evaluate this outcome measure of by looking at multiple variables indicating completion of target exercise. One of the variables used to assess this primary outcome measure of adherence is a summary of the Exercise Enjoyment Scale ratings of exercises to compare the study groups. This data will be extracted from the 7 Movements App.

SECONDARY OUTCOMES:
Qualitative Study Review; perceived acceptability of the intervention using a descriptive, open-ended questionnaire. | 12 weeks
  A qualitative study review to be done in partnership with participants upon completion. This outcome measure will be evaluated using a Post Intervention Descriptive Questionnaire to be completed by participants. Open-ended questions in this questionnaire will be cover 4 major themes. One of these themes is participants perceived acceptability of the intervention.
Qualitative Study Review; the identification of barriers or facilitators to the study using a descriptive, open-ended questionnaire. | 12 weeks
  A qualitative study review to be done in partnership with participants upon completion. This outcome measure will be evaluated using a Post Intervention Descriptive Questionnaire to be completed by participants. Open-ended questions in this questionnaire will be cover 4 major themes. One of these themes is participants identification of barriers and facilitators to study activity.
Qualitative Study Review; participant assessment of the 7 Movements App and technology using a descriptive, open-ended questionnaire. | 12 weeks
  A qualitative study review to be done in partnership with participants upon completion. This outcome measure will be evaluated using a Post Intervention Descriptive Questionnaire to be completed by participants. Open-ended questions in this questionnaire will be cover 4 major themes. One of these themes is participants opinions of the 7 Movements platform and technology.
Qualitative Study Review; study safety concerns as expressed by participants using a descriptive, open-ended questionnaire. | 12 weeks
  A qualitative study review to be done in partnership with participants upon completion. This outcome measure will be evaluated using a Post Intervention Descriptive Questionnaire to be completed by participants. Open-ended questions in this questionnaire will be cover 4 major themes. One of these themes is adverse events or safety concerns, as expressed by participants.
Actigraphy: heart rate measures (bpm). | 12 weeks
  Actigraphy data (segmented as sedentary time or mild/moderate/vigorous activity) from five day windows pre-study and post-study. Data collected will include heart rate data collected during two 5 day windows within the study period to assess the effect of Exercise Snack and active movement break interventions on heart rate. The Actigraph LEAP measures heart rate (bpm) using a photoplethysmography (PPG) sensor, a common technology for non-invasive heart rate monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Daryl J Wile, MD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia Okanagan, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with our Collaborators:
  Dr. Jonathan Little, Health and Exercise Sciences, UBCO, primary research focus is on how the application of different nutrition and exercise strategies impact glucose control, cardiometabolic health, and inflammation. Dr. Little specializes in the use of exercise snacks for health interventions.
  Dr. Mary Jung - Health and Exercise Science, UBCO, primary research focus is in health promotion and health behavior changes.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: April 1, 2025 until study completion
Access Criteria: Only those listed on the approved REB application will have access to IPD.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-03-11): https://cdn.clinicaltrials.gov/large-docs/87/NCT06915987/Prot_SAP_000.pdf
  • Informed Consent Form (2025-03-11): https://cdn.clinicaltrials.gov/large-docs/87/NCT06915987/ICF_001.pdf